CLINICAL TRIAL: NCT02918266
Title: A Randomized, Double-Blind, Sponsor Unblinded, Placebo-Controlled, 5-Period Crossover, Phase 1b Study To Evaluate The Effects Of Single Oral Administration of TAK-071 On Scopolamine-Induced Cognitive Impairment In Healthy Subjects
Brief Title: TAK-071 Scopolamine-Induced Cognitive Impairment Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated prematurely due to indication change.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: TAK-071-1002; U1111-1184-2278 (Registry Identifier: WHO)
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — Scopolamine; TAK-071; Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (11):
- Part 1: TAK-071 80 mg + Scopolamine 0.5 mg (Experimental): TAK-071 80 milligram (mg), drug in capsule (DIC), orally, Day 1, followed by scopolamine 0.5 mg, injection, subcutaneously, Day 2. TAK-071 will be taken 24 hours before scopolamine injection.
  Interventions: Drug: Scopolamine; Drug: TAK-071
- Part 2: Treatment Sequence ABDEC (Experimental): TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection,SC,Day2 of Period1(A); followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period2(B);followed by TAK-071 80mg, DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period3(D);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period4(E);followed by TAK-071 80mg, DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period5(C). TAK-071 and donepezil will be taken 24 and 3 hours before scopolamine injection. A washout period of 3-weeks will be maintained between each treatment period.
  Interventions: Drug: Scopolamine; Drug: TAK-071; Drug: Donepezil; Drug: Scopolamine Placebo; Drug: TAK-071 Placebo; Drug: Donepezil Placebo
- Part 2: Treatment Sequence BCEAD (Experimental): TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period1(B);followed by TAK-071 80mg, DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period2(C);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period3(E);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection,SC,Day2 of Period4(A);followed by TAK-071 80mg, DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period5(D). TAK-071 and donepezil will be taken 24 and 3 hours before scopolamine injection. A washout period of 3-weeks will be maintained between each treatment period.
  Interventions: Drug: Scopolamine; Drug: TAK-071; Drug: Donepezil; Drug: Scopolamine Placebo; Drug: TAK-071 Placebo; Drug: Donepezil Placebo
- Part 2: Treatment Sequence CDABE (Experimental): TAK-071 80mg, DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period1(C);followed by TAK-071 80mg, DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period2(D);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection,SC,Day2 of Period3(A);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period4(B);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period5(E). TAK-071 and donepezil will be taken 24 and 3 hours before scopolamine injection. A washout period of 3-weeks will be maintained between each treatment period.
  Interventions: Drug: Scopolamine; Drug: TAK-071; Drug: Donepezil; Drug: Scopolamine Placebo; Drug: TAK-071 Placebo; Drug: Donepezil Placebo
- Part 2: Treatment Sequence DEBCA (Experimental): TAK-071 80mg, DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period1(D);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period2(E);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period3(B);followed by TAK-071 80mg, DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period4(C);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection,SC,Day2 of Period5(A). TAK-071 and donepezil will be taken 24 and 3 hours before scopolamine injection. A washout period of 3-weeks will be maintained between each treatment period.
  Interventions: Drug: Scopolamine; Drug: TAK-071; Drug: Donepezil; Drug: Scopolamine Placebo; Drug: TAK-071 Placebo; Drug: Donepezil Placebo
- Part 2: Treatment Sequence EACDB (Experimental): TAK-071 placebo-matching DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period1(E);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection,SC,Day2 of Period2(A);followed by TAK-071 80mg, DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period3(C);followed by TAK-071 80mg, DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period4(D);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period5(B). TAK-071 and donepezil will be taken 24 and 3 hours before scopolamine injection. A washout period of 3-weeks will be maintained between each treatment period.
  Interventions: Drug: Scopolamine; Drug: TAK-071; Drug: Donepezil; Drug: Scopolamine Placebo; Drug: TAK-071 Placebo; Drug: Donepezil Placebo
- Part 2: Treatment Sequence ACBED (Experimental): TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection,SC,Day2 of Period1(A);followed by TAK-071 80mg, DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period2(C);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period3(B);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period4(E);followed by TAK-071 80mg, DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period5(D). TAK-071 and donepezil will be taken 24 and 3 hours before scopolamine injection. A washout period of 3-weeks will be maintained between each treatment period.
  Interventions: Drug: Scopolamine; Drug: TAK-071; Drug: Donepezil; Drug: Scopolamine Placebo; Drug: TAK-071 Placebo; Drug: Donepezil Placebo
- Part 2: Treatment Sequence BDCAE (Experimental): TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period1(B);followed by TAK-071 80mg, DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period2(D);followed by TAK-071 80mg, DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period3(C);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection,SC,Day2 of Period4(A);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period5(E). TAK-071 and donepezil will be taken 24 and 3 hours before scopolamine injection. A washout period of 3-weeks will be maintained between each treatment period.
  Interventions: Drug: Scopolamine; Drug: TAK-071; Drug: Donepezil; Drug: Scopolamine Placebo; Drug: TAK-071 Placebo; Drug: Donepezil Placebo
- Part 2: Treatment Sequence CEDBA (Experimental): TAK-071 80mg, DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period1(C);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period2(E);followed by TAK-071 80mg, DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period3(D);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period4(B);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection,SC,Day2 of Period5(A). TAK-071 and donepezil will be taken 24 and 3 hours before scopolamine injection. A washout period of 3-weeks will be maintained between each treatment period.
  Interventions: Drug: Scopolamine; Drug: TAK-071; Drug: Donepezil; Drug: Scopolamine Placebo; Drug: TAK-071 Placebo; Drug: Donepezil Placebo
- Part 2: Treatment Sequence DAECB (Experimental): TAK-071 80mg, DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period1(D);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection,SC,Day2 of Period2(A);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period3(E);followed by TAK-071 80mg, DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period4(C); followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period5(B). TAK-071 and donepezil will be taken 24 and 3 hours before scopolamine injection. A washout period of 3-weeks will be maintained between each treatment period.
  Interventions: Drug: Scopolamine; Drug: TAK-071; Drug: Donepezil; Drug: Scopolamine Placebo; Drug: TAK-071 Placebo; Drug: Donepezil Placebo
- Part 2: Treatment Sequence EBADC (Experimental): TAK-071 placebo-matching DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period1(E);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period2(B);followed by TAK-071 placebo-matching DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection,SC,Day2 of Period3(A);followed by TAK-071 80mg, DIC, orally,Day1, donepezil 10mg, over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period4(D);followed by TAK-071 80mg, DIC, orally,Day1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5mg, injection,SC,Day2 of Period5(C). TAK-071 and donepezil will be taken 24 and 3 hours before scopolamine injection. A washout period of 3-weeks will be maintained between each treatment period.
  Interventions: Drug: Scopolamine; Drug: TAK-071; Drug: Donepezil; Drug: Scopolamine Placebo; Drug: TAK-071 Placebo; Drug: Donepezil Placebo

INTERVENTIONS:
Drug: Scopolamine — Scopolamine subcutaneous injection
Drug: TAK-071 — TAK-071 DIC
Drug: Donepezil — Donepezil over-encapsulated tablet
  Arms: Part 2: Treatment Sequence ABDEC; Part 2: Treatment Sequence ACBED; Part 2: Treatment Sequence BCEAD; Part 2: Treatment Sequence BDCAE; Part 2: Treatment Sequence CDABE; Part 2: Treatment Sequence CEDBA; Part 2: Treatment Sequence DAECB; Part 2: Treatment Sequence DEBCA; Part 2: Treatment Sequence EACDB; Part 2: Treatment Sequence EBADC
Drug: Scopolamine Placebo — Scopolamine placebo-matching subcutaneous injection
  Arms: Part 2: Treatment Sequence ABDEC; Part 2: Treatment Sequence ACBED; Part 2: Treatment Sequence BCEAD; Part 2: Treatment Sequence BDCAE; Part 2: Treatment Sequence CDABE; Part 2: Treatment Sequence CEDBA; Part 2: Treatment Sequence DAECB; Part 2: Treatment Sequence DEBCA; Part 2: Treatment Sequence EACDB; Part 2: Treatment Sequence EBADC
Drug: TAK-071 Placebo — TAK-071 placebo-matching DIC
  Arms: Part 2: Treatment Sequence ABDEC; Part 2: Treatment Sequence ACBED; Part 2: Treatment Sequence BCEAD; Part 2: Treatment Sequence BDCAE; Part 2: Treatment Sequence CDABE; Part 2: Treatment Sequence CEDBA; Part 2: Treatment Sequence DAECB; Part 2: Treatment Sequence DEBCA; Part 2: Treatment Sequence EACDB; Part 2: Treatment Sequence EBADC
Drug: Donepezil Placebo — Donepezil placebo-matching over-encapsulated tablet
  Arms: Part 2: Treatment Sequence ABDEC; Part 2: Treatment Sequence ACBED; Part 2: Treatment Sequence BCEAD; Part 2: Treatment Sequence BDCAE; Part 2: Treatment Sequence CDABE; Part 2: Treatment Sequence CEDBA; Part 2: Treatment Sequence DAECB; Part 2: Treatment Sequence DEBCA; Part 2: Treatment Sequence EACDB; Part 2: Treatment Sequence EBADC

SUMMARY:
The purpose of this study is to assess the effect of a single oral dose of TAK-071 on the attenuation of cognitive deficit induced by scopolamine as measured by Groton Maze Learning Test (GMLT) (total number of errors).

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-071. This study will look at the effect of a single oral dose of TAK-071, a novel muscarinic acetylcholine receptor 1 positive allosteric modulator, on scopolamine-induced deficits in cognitive function in healthy adult male participants. The study consists of two parts: Part 1 is a substudy to explore PK profile of TAK-071 in the presence of light meal and coadministration of scopolamine to determine TAK-071 dose for the next part; Part 2 is the main the study to assess the effects of TAK-071 on scopolamine-induced cognitive impairment. The study will enroll approximately 6 participants in Part 1 and 40 participants in Part 2. Participant will be assigned to received TAK-071 along with scopolamine in Part 1 and will be randomly assigned to one of the ten treatment sequences in Part 2-which will remain undisclosed to the participants and study doctor during the study (unless there is an urgent medical need):

Part 2: Treatment Sequence ABDEC Part 2: Treatment Sequence BCEAD Part 2: Treatment Sequence CDABE Part 2: Treatment Sequence DEBCA Part 2: Treatment Sequence EACDB Part 2: Treatment Sequence ACBED Part 2: Treatment Sequence BDCAE Part 2: Treatment Sequence CEDBA Part 2: Treatment Sequence DAECB Part 2: Treatment Sequence EBADC Where A=scopolamine matching placebo SC + TAK-071 matching placebo oral (PO) + donepezil matching placebo PO; B=scopolamine 0.5 mg SC + TAK-071 matching placebo PO + donepezil matching placebo PO; C=scopolamine 0.5 mg SC + TAK-071 PO + donepezil matching placebo PO; D=scopolamine 0.5 mg SC + TAK-071 PO + donepezil 10 mg PO; and E=scopolamine 0.5 mg SC + TAK-071 matching placebo PO + donepezil 10 mg PO.

The dose of TAK-071 that was well-tolerated in the TAK-071-1001 study (NCT02769065) will be selected, based on the safety and tolerability data from the single-rising dose (SRD) study for administration in Part 1. Each participant will also receive scopolamine 0.5 mg, injection, SC, once at the time of Screening. This single center trial will be conducted in the United States. The overall time to participate in this study is approximately 5.7 weeks in Part 1 and 21 weeks in Part 2. Participants will remain confined to the clinic for 4 days during Part 1 and 3 days during the each intervention period in Part 2. Participants will be contacted by telephone on Day 12 in Part 1 and Day 9 of Period 5 in Part 2 for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Weighs at least 50 kilogram (kg) and has a body mass index (BMI) from 18.0 to 30.0 kilogram per square meter (kg/m^2), inclusive at Screening.

Additional inclusion criteria for Part 2:

1. Able to perform the CogState battery.
2. Change from Baseline (average) in total GMLT errors of less than or equal to (<=) -5 at 2 hours postdose of scopolamine.
3. Sleepiness score less than (<) 8 on the karolinska sleepiness scale (KSS) at 2 hours postdose of scopolamine.
4. Passes a hearing test with at least 80 percent (%) correct responses and no more than 20% false positives. This test can be repeated once to determine eligibility.

Exclusion Criteria:

1. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as regular consumption of 4 or more units per day) within 1 year prior to the Screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study. One unit is equivalent to a half-pint of beer or 1 measure of spirits or 1 glass of wine.
2. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in Day -1 of Period 1. Cotinine test is positive at Screening or Check-in (Day -1) of Period 1.
3. Has poor peripheral venous access.
4. Has donated or lost 450 milliliter (mL) or more of his blood volume (including plasmapheresis), or had a transfusion of any blood product within 30 days prior to Day 1 of Period 1.
5. Is a shift worker (night, late, or early resulting in irregular bed times) or has crossed or will cross more than 2 time zones within 48 hours in the period from 48 hours prior to Treatment Period 1, Day 1 until the end of Treatment Period 5.
6. Reports symptoms suggesting evidence of a current sleep disorder or history of sleep disorder, including but not limited to sleep apnea, heavy snoring, primary or chronic insomnia, narcolepsy or restless leg syndrome, as judged by medical history.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-11-21; Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United states from 21 November 2016 to 08 August 2017.
Pre-assignment Details: Healthy male participants were enrolled in this 2-part study to receive: TAK-071, scopolamine in Part 1; TAK-071, scopolamine and donepezil in a cross-over sequence in Part 2. The study was terminated prior to start of Part 2 intervention period 2 due to indication change.
Groups:
- Part 1: TAK-071 80 mg + Scopolamine 0.5 mg: TAK-071 80 milligram (mg), drug in capsule (DIC), orally, on Day 1, followed by scopolamine 0.5 mg, injection, subcutaneously (SC), on Day 2.
- Part 2: Treatment Sequence ABDEC: TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection, SC, on Day 2 of Period 1 (A); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 2 (B); followed by TAK-071 80 mg, DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 3 (D); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 4 (E); followed by TAK-071, DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 5 (C). A washout period of 3-weeks was maintained between each treatment period.
- Part 2: Treatment Sequence BCEAD: TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 1 (B); followed by TAK-071 80 mg, DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 2 (C); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 3 (E); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection, SC, on Day 2 of Period 4 (A); followed by TAK-071 80 mg, DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 5 (D). A washout period of 3-weeks was maintained between each treatment period.
- Part 2: Treatment Sequence CDABE: TAK-071 80 mg, DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 1 (C); followed by TAK-071 80 mg, DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 2 (D); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection, SC, on Day 2 of Period 3 (A); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 4 (B); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 5 (E). A washout period of 3-weeks was maintained between each treatment period
- Part 2: Treatment Sequence DEBCA: TAK-071 80 mg, DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 1 (D); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 2 (E); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 3 (B); followed by TAK-071 80 mg, DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 4 (C); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection, SC, on Day 2 of Period 5 (A). A washout period of 3-weeks was maintained between each treatment period.
- Part 2: Treatment Sequence EACDB: TAK-071 placebo-matching DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 1 (E); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection, SC, on Day 2 of Period 2 (A);followed by TAK-071 80 mg, DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 3 (C); followed by TAK-071 80 mg, DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 4 (D); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 5 (B). A washout period of 3-weeks was maintained between each treatment period.
- Part 2: Treatment Sequence ACBED: TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection, SC, on Day 2 of Period 1 (A); followed by TAK-071 DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 2 (C); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 3 (B); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 4 (E); followed by TAK-071 80 mg, DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 5 (D). A washout period of 3-weeks was maintained between each treatment period.
- Part 2: Treatment Sequence BDCAE: TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 1 (B);followed by TAK-071 80 mg, DIC, orally, Day1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 2 (D);followed by TAK-071 80 mg, DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 3 (C);followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection, SC, on Day 2 of Period 4 (A); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 5 (E). A washout period of 3-weeks was maintained between each treatment period.
- Part 2: Treatment Sequence CEDBA: TAK-071 80 mg, DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 1 (C); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 2 (E); followed by TAK-071 80 mg, DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 3 (D); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, Day 2 of Period 4 (B); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection, SC, on Day 2 of Period 5 (A). A washout period of 3-weeks was maintained between each treatment period.
- Part 2: Treatment Sequence DAECB: TAK-071 80 mg, DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 1 (D); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection, SC, on Day 2 of Period 2 (A); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 3 (E); followed by TAK-071 80 mg, DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 4 (C); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 5 (B). A washout period of 3-weeks was maintained between each treatment period.
- Part 2: Treatment Sequence EBADC: TAK-071 80 mg, placebo-matching DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 1 (E); followed by TAK-071 placebo-matching DIC, orally, Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 2 (B); followed by TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection, SC, on Day 2 of Period 3 (A); followed by TAK-071 80 mg, DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 4 (D); followed by TAK-071 80 mg, DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 of Period 5 (C). A washout period of 3-weeks was maintained between each treatment period.
Period: Part 1
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment Sequence ABDEC | Part 2: Treatment Sequence BCEAD | Part 2: Treatment Sequence CDABE | Part 2: Treatment Sequence DEBCA | Part 2: Treatment Sequence EACDB | Part 2: Treatment Sequence ACBED | Part 2: Treatment Sequence BDCAE | Part 2: Treatment Sequence CEDBA | Part 2: Treatment Sequence DAECB | Part 2: Treatment Sequence EBADC
Started | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Intervention Period 1 (2 Days)
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment Sequence ABDEC | Part 2: Treatment Sequence BCEAD | Part 2: Treatment Sequence CDABE | Part 2: Treatment Sequence DEBCA | Part 2: Treatment Sequence EACDB | Part 2: Treatment Sequence ACBED | Part 2: Treatment Sequence BDCAE | Part 2: Treatment Sequence CEDBA | Part 2: Treatment Sequence DAECB | Part 2: Treatment Sequence EBADC
Started | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 1
Not completed — Study termination | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 1
Period: Part 2: Washout Period 1 (3 Weeks)
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment Sequence ABDEC | Part 2: Treatment Sequence BCEAD | Part 2: Treatment Sequence CDABE | Part 2: Treatment Sequence DEBCA | Part 2: Treatment Sequence EACDB | Part 2: Treatment Sequence ACBED | Part 2: Treatment Sequence BDCAE | Part 2: Treatment Sequence CEDBA | Part 2: Treatment Sequence DAECB | Part 2: Treatment Sequence EBADC
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Intervention Period 2 (2 Days)
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment Sequence ABDEC | Part 2: Treatment Sequence BCEAD | Part 2: Treatment Sequence CDABE | Part 2: Treatment Sequence DEBCA | Part 2: Treatment Sequence EACDB | Part 2: Treatment Sequence ACBED | Part 2: Treatment Sequence BDCAE | Part 2: Treatment Sequence CEDBA | Part 2: Treatment Sequence DAECB | Part 2: Treatment Sequence EBADC
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Washout Period 2 (3 Weeks)
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment Sequence ABDEC | Part 2: Treatment Sequence BCEAD | Part 2: Treatment Sequence CDABE | Part 2: Treatment Sequence DEBCA | Part 2: Treatment Sequence EACDB | Part 2: Treatment Sequence ACBED | Part 2: Treatment Sequence BDCAE | Part 2: Treatment Sequence CEDBA | Part 2: Treatment Sequence DAECB | Part 2: Treatment Sequence EBADC
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Intervention Period 3 (2 Days)
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment Sequence ABDEC | Part 2: Treatment Sequence BCEAD | Part 2: Treatment Sequence CDABE | Part 2: Treatment Sequence DEBCA | Part 2: Treatment Sequence EACDB | Part 2: Treatment Sequence ACBED | Part 2: Treatment Sequence BDCAE | Part 2: Treatment Sequence CEDBA | Part 2: Treatment Sequence DAECB | Part 2: Treatment Sequence EBADC
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Washout Period 3 (3 Weeks)
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment Sequence ABDEC | Part 2: Treatment Sequence BCEAD | Part 2: Treatment Sequence CDABE | Part 2: Treatment Sequence DEBCA | Part 2: Treatment Sequence EACDB | Part 2: Treatment Sequence ACBED | Part 2: Treatment Sequence BDCAE | Part 2: Treatment Sequence CEDBA | Part 2: Treatment Sequence DAECB | Part 2: Treatment Sequence EBADC
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Intervention Period 4 (2 Days)
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment Sequence ABDEC | Part 2: Treatment Sequence BCEAD | Part 2: Treatment Sequence CDABE | Part 2: Treatment Sequence DEBCA | Part 2: Treatment Sequence EACDB | Part 2: Treatment Sequence ACBED | Part 2: Treatment Sequence BDCAE | Part 2: Treatment Sequence CEDBA | Part 2: Treatment Sequence DAECB | Part 2: Treatment Sequence EBADC
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Washout Period 4 (3 Weeks)
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment Sequence ABDEC | Part 2: Treatment Sequence BCEAD | Part 2: Treatment Sequence CDABE | Part 2: Treatment Sequence DEBCA | Part 2: Treatment Sequence EACDB | Part 2: Treatment Sequence ACBED | Part 2: Treatment Sequence BDCAE | Part 2: Treatment Sequence CEDBA | Part 2: Treatment Sequence DAECB | Part 2: Treatment Sequence EBADC
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2: Intervention Period 5 (2 Days)
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment Sequence ABDEC | Part 2: Treatment Sequence BCEAD | Part 2: Treatment Sequence CDABE | Part 2: Treatment Sequence DEBCA | Part 2: Treatment Sequence EACDB | Part 2: Treatment Sequence ACBED | Part 2: Treatment Sequence BDCAE | Part 2: Treatment Sequence CEDBA | Part 2: Treatment Sequence DAECB | Part 2: Treatment Sequence EBADC
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were enrolled and received 1 dose of study drug.
Groups:
- Part 1: TAK-071 80 mg + Scopolamine 0.5 mg: TAK-071 80 mg, DIC, orally, on Day 1, followed by scopolamine 0.5 mg, injection, SC, on Day 2. TAK-071 will be taken 24 hours before scopolamine injection.
- Total: Total of all reporting groups
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment Sequence ABDEC | Part 2: Treatment Sequence BCEAD | Part 2: Treatment Sequence CDABE | Part 2: Treatment Sequence DEBCA | Part 2: Treatment Sequence EACDB | Part 2: Treatment Sequence ACBED | Part 2: Treatment Sequence BDCAE | Part 2: Treatment Sequence CEDBA | Part 2: Treatment Sequence DAECB | Part 2: Treatment Sequence EBADC | Total
Number analyzed (Participants) | 6 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 18
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 8
  Not Hispanic or Latino | 3 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 5
  White | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 10
  More than one race | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 18
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 6 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 1 | 0 | 16
  Current smoker | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ex-smoker | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Alcohol Classification [Count of Participants; unit: Participants]
  Never drunk | 3 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 10
  Current drinker: had less than (<) 4 units per day | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 7
  Current drinker: had 4 or more units per day | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ex-drinker | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Caffeine Consumption [Count of Participants; unit: Participants]
  Had caffeine consumption | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 5
  Had no caffeine consumption | 4 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 13
Academic Qualifications [Count of Participants; unit: Participants]
  No degree or diploma | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Elementary school | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  High school | 3 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 6
  Non university degree | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  University | 3 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Part 2: Change From Baseline in Total Number of Errors on the Groton Maze Learning Test (GMLT) at 2 Hours Post-Scopolamine Dose on Day 2
Time Frame: Baseline, 2 hours post scopolamine dose on Day 2
Population: No data was collected for Part 2 due to premature study termination because of indication change.
Groups:
- Part 2: Treatment A: TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine placebo-matching injection, SC, on Day 2 in each intervention period.
- Part 2: Treatment B: TAK-071 placebo-matching DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 in each intervention period.
- Part 2: Treatment C: TAK-071 80 mg, DIC, orally, on Day 1, donepezil placebo-matching over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 in each intervention period.
- Part 2: Treatment D: TAK-071 80 mg, DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 in each intervention period.
- Part 2: Treatment E: TAK-071 placebo-matching DIC, orally, on Day 1, donepezil 10 mg, over-encapsulated tablet, orally along with scopolamine 0.5 mg, injection, SC, on Day 2 in each intervention period.
Arm/Group | Part 2: Treatment A | Part 2: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Part 2: Treatment E
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Part 2: Change From Baseline in Total Number of Errors on the GMLT
Time Frame: Baseline, Day 2 at multiple time points post-scopolamine dose (up to 10 hours)
Population: No data was collected for Part 2 due to premature study termination because of indication change.
Arm/Group | Part 2: Treatment A | Part 2: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Part 2: Treatment E
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Part 2: AUECt: GMLT Area Under the Effect Curve From Time 0 Hours to Time t (AUECt) (Net Area) for TAK-071
Time Frame: Day 2 pre-dose and at multiple time points (up to 10 hours) post-scopolamine dose
Population: No data was collected for Part 2 due to premature study termination because of indication change.
Arm/Group | Part 2: Treatment A | Part 2: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Part 2: Treatment E
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Part 2: Emax: GMLT Maximum Observed Effect (Emax) for TAK-071
Time Frame: Day 2 pre-dose and at multiple time points (up to 10 hours) post-scopolamine dose
Population: No data was collected for Part 2 due to premature study termination because of indication change.
Arm/Group | Part 2: Treatment A | Part 2: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Part 2: Treatment E
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Part 2: TEmax: Time to Reach GMLT Emax for TAK-071
Time Frame: Day 2 pre-dose and at multiple timepoints (up to 10 hours) post-scopolamine dose
Population: No data was collected for Part 2 due to premature study termination because of indication change.
Arm/Group | Part 2: Treatment A | Part 2: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Part 2: Treatment E
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants Who Experienced at Least One Treatment-emergent Adverse Event (TEAE)
Time Frame: Part 1: Baseline up to Day 12; Part 2: Baseline up to Day 9 of Period 1
Population: The safety analysis set included all participants who were enrolled and received 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Scopolamine 0.5 mg SC + TAK-071 80 mg: TAK-071 80 mg, DIC, orally, on Day 1, followed by scopolamine 0.5 mg, injection, subcutaneously, on Day 2. TAK-071 will be taken 24 hours before scopolamine injection.
Arm/Group | Scopolamine 0.5 mg SC + TAK-071 80 mg | Part 2: Treatment A | Part 2: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Part 2: Treatment E
Number analyzed (Participants) | 6 | 3 | 2 | 3 | 2 | 2
percentage of participants | 66.7 | 66.7 | 100.0 | 100.0 | 100.0 | 100.0

7. Secondary Outcome: Percentage of Participants Who Meet the Takeda Markedly Abnormal Criteria for Clinical Laboratory Tests at Least Once Postdose
Time Frame: Part 1: Baseline up to Day 12; Part 2: Baseline up to Day 9 of Period 1
Population: The safety analysis set included all participants who were enrolled and received 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Scopolamine 0.5 mg SC + TAK-071 80 mg | Part 2: Treatment A | Part 2: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Part 2: Treatment E
Number analyzed (Participants) | 6 | 3 | 2 | 3 | 2 | 2
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants Who Meet the Takeda Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Postdose
Time Frame: Part 1: Baseline up to Day 12; Part 2: Baseline up to Day 9 of Period 1
Population: The safety analysis set included all participants who were enrolled and received 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment A | Part 2: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Part 2: Treatment E
Number analyzed (Participants) | 6 | 3 | 2 | 3 | 2 | 2
percentage of participants
  Diastolic Blood Pressure (mmHg)/Supine <50 mmHg | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate/supine: <50 beats per minute | 33.3 | 33.3 | 50.0 | 0 | 0 | 50.0
  Temperature: <35.6 Celsius | 0 | 0 | 0 | 33.3 | 0 | 0
  Temperature: >37.7 Celsius | 16.7 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Percentage of Participants Who Meet the Takeda Markedly Abnormal Criteria for Electrocardiogram (ECG) at Least Once Postdose
Time Frame: Part 1: Baseline up to Day 12; Part 2: Baseline up to Day 9 of Period 1
Population: The safety analysis set included all participants who were enrolled and received 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment A | Part 2: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Part 2: Treatment E
Number analyzed (Participants) | 6 | 3 | 2 | 3 | 2 | 2
percentage of participants | 16.7 | 0 | 50.0 | 0 | 0 | 50.0

10. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-071
Time Frame: Part 1: Day 1 pre-TAK-071 dose and at multiple time points (up to 168 hours) post-TAK-071 dose; Part 2: Day 2 pre-TAK-071 dose and at multiple time points (up to 10 hours) post-scopolamine dose
Population: The pharmacokinetic (PK) set included all participants who received study drug and had at least 1 measurable plasma concentration. No data was collected for Part 2 due to premature study termination because of indication change.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment A | Part 2: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Part 2: Treatment E
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0
nanogram per milliliter (ng/mL) | 1066 (16.8) |  |  |  |  |

11. Secondary Outcome: Tmax: Time to Reach the Maximum Observed Plasma Concentration(Cmax) for TAK-071
Time Frame: as for outcome 10
Population: The PK set included all participants who received study drug and had at least 1 measurable plasma concentration. No data was collected for Part 2 due to premature study termination because of indication change.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment A | Part 2: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Part 2: Treatment E
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0
hours | 30.00 [12.0 to 34.0] |  |  |  |  |

12. Secondary Outcome: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-071
Time Frame: as for outcome 10
Population: The PK set included all participants who received study drug and had at least 1 measurable plasma concentration.No data was collected for Part 2 due to premature study termination because of indication change.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment A | Part 2: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Part 2: Treatment E
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0
hour*nanogram per milliliter (h*ng/mL) | 82010 (25.0) |  |  |  |  |

13. Secondary Outcome: AUC24: Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours Postdose for TAK-071
Time Frame: Part 1: Day 1 pre-TAK-071 dose and at multiple time points (up to 24 hours) post-TAK-071 dose; Part 2: Day 2 pre-TAK-071 dose and at multiple time points (up to 24 hours) post-scopolamine dose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment A | Part 2: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Part 2: Treatment E
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0
h*ng/mL | 19330 (16.0) |  |  |  |  |

14. Secondary Outcome: AUCt1-t2: Area Under the Plasma Concentration-Time Curve From Time t1 to Time t2 for TAK-071
Time Frame: as for outcome 10
Population: As per change in planned analyses, data was not collected.
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment A | Part 2: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Part 2: Treatment E
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: AUC∞: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity for TAK-071
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment A | Part 2: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Part 2: Treatment E
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0
h*ng/mL | 94100 (26.8) |  |  |  |  |

16. Secondary Outcome: T1/2z: Terminal Disposition Phase Elimination Half-Life in Plasma for TAK-071
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment A | Part 2: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Part 2: Treatment E
Number analyzed (Participants) | 6 | 0 | 0 | 0 | 0 | 0
hours | 47.02 (14.864) |  |  |  |  |

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) are adverse events that started after the first dose of study drug up to Day 12 in Part 1 and Day 9 of Period 1 in Part 2 (study termination) after the last dose of study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg | Part 2: Treatment A | Part 2: Treatment B | Part 2: Treatment C | Part 2: Treatment D | Part 2: Treatment E
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/2 | 0/3 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/2 | 0/3 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 4/6 | 2/3 | 2/2 | 3/3 | 2/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: TAK-071 80 mg + Scopolamine 0.5 mg (N=6) | Part 2: Treatment A (N=3) | Part 2: Treatment B (N=2) | Part 2: Treatment C (N=3) | Part 2: Treatment D (N=2) | Part 2: Treatment E (N=2)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 4 | 2 | 1 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT02918266/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/66/NCT02918266/SAP_001.pdf